CLINICAL TRIAL: NCT05299255
Title: An Open, Single-center Phase II Clinical Study of Utidelone in Third-line and Above Treatment of Small Cell Lung Cancer
Brief Title: Utidelone in Third-line and Above Treatment of Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Yanqiu Zhao, Head of Oncology, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HXNI-YTDL-001
Record Dates: First submitted 2022-03-08; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: SCLC, Extensive Stage
Keywords: small cell lung cancer,Utidelone
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Utidelone vs placebo (Experimental): Drug: Utidelone vs placebo in Third-line and above Treatment Extensive Small-cell Lung Cancer
  Interventions: Drug: Utidelone; Drug: Placebo

INTERVENTIONS:
Drug: Utidelone — Utidelone Versus placebo in Third-line and above treatment of Extensive Small-cell Lung Cancer
Drug: Placebo — the placebo as control group.

SUMMARY:
SCLC has a very high degree of malignancy, and 60% to 70% of patients are diagnosed as extensive stage. The median survival of patients with limited-stage disease is about 15-20 months, and the median OS of patients with extensive-stage disease is about 8-13 months, and the 2-year and 5-year survival rates are about 5% and 1-2%, respectively. However, although the initial treatment has a high effective rate, most patients relapse or progress within 1 year, and the effect of re-treatment is poor and the prognosis is poor. The effective rate of SCLC second-line treatment is only 10-25%, and the median survival time is less than 6 months. After the third and fourth lines, there are almost no recognized treatment options. Therefore, improving the second-line treatment of SCLC has always been a difficult clinical problem, and new drugs are urgently needed to be explored. In small cell lung cancer, based on phase II clinical trials, paclitaxel is currently recommended by NCCN guidelines for subsequent systemic therapy in patients who relapse 6 months or less after initial therapy. Utidelone (UTD1) is an epothilone derivative with a similar mechanism of action to taxanes, but a completely different molecular structure.

DETAILED DESCRIPTION:
Compared with paclitaxel, epothilones has higher water solubility and toxicity tolerance, and fewer side effects, these findings suggest that utidron may have better antitumor activity against small cell lung cancer. Therefore, to prospectively observe the treatment of extensive-stage small cell lung cancer with failure of second-line or above chemotherapy and receive Utilidron, so as to understand the efficacy, safety and tolerability of Utilidron in the third-line and above treatment of small cell lung cancer, which is a small Post-line treatment of cell lung cancer provides new directions and treatment options.

This study is an open, single-center phase II clinical study. Small cell lung cancer patients with disease progression or recurrence after second-line therapy or above, receive Utilidron injection. Utilidron injection 40mg/m2/d d1-5 q3w was administered until disease progression (PD), intolerable toxicity, initiation of new antitumor therapy, loss to follow-up, death, and the investigator decided to be tested Subjects who withdraw from the study treatment or the subject/their legal representative requests to withdraw from the study (whichever occurs first). After consultation with the sponsor, the patient will determine whether the treatment can be continued, observe and evaluate the preliminary efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed small cell lung cancer (except for small cell lung cancer mixed with other pathological types);
* The expected survival period is not less than 3 months;
* Second-line therapy (excluding maintenance therapy) and above with disease progression or recurrence of small cell lung cancer;
* Patients who have not received chemotherapy, radiotherapy, surgery, targeted therapy and immunotherapy within 4 weeks before enrollment;
* Age 18-75 years old, physical condition score ECOG 0-1 points;
* At least one target lesion measurable by imaging within 3 weeks before enrollment, ordinary CT scan ≥ 20 mm, spiral CT scan diameter ≥ 10 mm (lymph node short diameter ≥ 15 mm);
* Asymptomatic brain metastases, or patients with stable disease for more than 4 weeks after brain metastases treatment;
* Neurological lesions should be less than grade 2 within 4 weeks before enrollment (NCI CTC4.03);
* Routine blood and blood biochemical tests were basically normal within 1 week before enrollment (based on the normal value of the research center laboratory, no blood transfusion within 14 days before screening, and no rhG-CSF was used):

Blood routine: HGB≥9g/dL; ANC≥1.5×109/L; PLT≥80×109/L; Blood biochemistry (without ALB infusion within 14 days): bilirubin <1.5 times the upper limit of normal, ALT and AST ≤2.5 times the upper limit of normal (if liver metastases exist, bilirubin ≤3 times the upper limit of normal, ALT and AST≤3 times the upper limit of normal) 5 times the upper limit of normal), serum Cr≤1.5 times the upper limit of normal or endogenous creatinine clearance ≥45 mL/min (Cockcroft-Gault formula);

* Those who have no major organ dysfunction and no concomitant heart disease;
* Females of childbearing age, including those who are in menopause but have not reached postmenopausal state (natural amenorrhea for 12 consecutive months) and who have not received sterilization and ovarian and/or hysterectomy, must have a blood pregnancy test within 7 days before the first

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or lactating patients;
* Patients with active pulmonary tuberculosis;
* Patients with high suspicion of interstitial lung disease;
* Exclusion criteria for combined diseases:

  * Cancerous meningitis patients;

    * patients with symptomatic central nervous system (CNS) metastasis;

      * Other active malignant tumors that require concurrent treatment, but not including carcinoma in situ of the cervix or basal cell carcinoma of the skin;

        * Patients with serious diseases, including severe heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, severe infection, active peptic ulcer, and those with a history of mental illness that is not easy to control;
* HIV positive test results, untreated active hepatitis patients;
* Patients with poor compliance; The investigators believe that those who are not suitable to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-05 (Actual); Primary Completion 2022-09-05 (Estimated); Study Completion 2023-09-05 (Estimated)

PRIMARY OUTCOMES:
The objective response rate (ORR) according to the RECIST 1.1 | 24 weeks
  the objective response rate (ORR）of utidelone in the third-Line and above treatment of ES-SCLC

CONTACTS AND LOCATIONS:
Overall Officials: Yanqiu Zhao, MS, Principal Investigator — Henan Tumor Hospital
Locations (1):
- Henan Tumor Hospital, Zhengzhou, Henan, China